CLINICAL TRIAL: NCT02007993
Title: Photodynamic Therapy as Novel Treatment for Halitosis in Adolescents: Crontolled Clinical Trial
Brief Title: Photodynamic Therapy in Adolescents Halitosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Rubia Garcia Lopes, master's degree student, University of Nove de Julho
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: halitose01
Record Dates: First submitted 2013-11-26; First posted 2013-12-11 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2013-12

CONDITIONS: Halitosis
Keywords: Halitosis,; Photodynamic Therapy,; Adolescent
MeSH Terms: conditions — Halitosis | interventions — 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 (Active Comparator): Treatment with a tongue scraper
  Interventions: Other: Tongue Scraper
- Group 2 (Experimental): PDT wavelength = 660 nm Fluency = 320 J/cm2 Power = 100 milliwatt Energy = 9 J Time = 90 s
  Interventions: Other: PDT
- Group 4 (Experimental): Tongue scraper + PDT wavelength = 660 nm Fluency = 320 J/cm2 Power = 100 milliwatt Energy = 9 J Time = 90 s
  Interventions: Other: PDT; Other: Tongue Scraper
- Group 3 (Experimental): PDT wavelength = 660 nm Fluency = 428 J/cm2 Power = 100 milliwatt Energy = 12 J Time = 120 s
  Interventions: Other: PDT
- Group 5 (Experimental): Tongue scraper + PDT wavelength = 660 nm Fluency = 428 J/cm2 Power = 100 milliwatt Energy = 12 J Time = 120 s
  Interventions: Other: PDT; Other: Tongue Scraper

INTERVENTIONS:
Other: PDT — A single session of PDT will be performed with the Chimiolux® photosensitizer at a concentration of 0.005% applied over the middle and posterior thirds of the dorsum of the tongue.
  Nine points will be irradiated, the device will be previously calibrated with a wavelength of 660 nm, power of 100 mW, energy of 9 joules for 90 seconds per point in Groups 2 and 4 and 12 joules for 120 second per point in Groups 3 and 5
  Arms: Group 2; Group 3; Group 4; Group 5
Other: Tongue Scraper — The pacient will scrap the tongue 10 times.
  Arms: Group 1; Group 4; Group 5

SUMMARY:
The aim of the proposed controlled clinical trial is to evaluate the effect of photodynamic therapy (PDT) on the formation of volatile sulfur compounds (VSCs) from coated tongue and its action on the severity of halitosis in adolescents using different treatment protocols.

HYPOTHESIS

1. - Null hypothesis: There is no change in halitosis following the use of photodynamic therapy.
2. - Experimental hypothesis: There is a reduction in halitosis following the use of photodynamic therapy alone or in combination with a tongue scraper.

DETAILED DESCRIPTION:
Halitosis (bad breath) is a term used to describe an unpleasant odor emanating from the mouth that could originate in the oral cavity itself or as a result of systemic factors. Halitosis is a common problem that affects most of the population worldwide and is caused mainly by the volatile sulfur compounds produced by anaerobic Gram-negative microorganisms in the oral cavity on sulfur-containing substrates in the oral cavity. On the dorsum of the tongue, the volatile sulfur compounds produced from this metabolism are hydrogen sulfide (H2S), methyl mercaptan (CH3SH3) and dimethyl sulfide (CH3-S-CH3). The concentration of these gases is used as an indicator of the severity of halitosis. Recently, the Gram positive anaerobic bacterium Solobacterium moorei (formerly known as Bulleidia moorei) has also been associated with oral malodor by volatile sulfur compounds production, particularly hydrogen sulfide in the presence of different supplements with amino acids more specifically cysteine, wich agrees with studies showing that the cysteine challenge is a in vivo and in vitro model for analyzing the production of hydrogen sulfide.

The measure of volatile sulfur compounds can be performed by an organoleptic evaluation of the air emanating from the oral cavity through gas chromatography or the use of a sulfide monitor, such at the Halimeter (Interscan Corporation), which determines the amount of volatile sulfur compounds in parts per billion (ppb) in the exhaled air. Gas chromatography is the most appropriate means for detecting halitosis of different origins. In 2004, the Oral ChromaTM (Abilit Corporation) was developed in Japan for the individual measurement of the three main gases (hydrogen sulfide, methyl mercaptan and dimethyl sulfide), allowing the evaluation of the intensity and origin of halitosis.

Light, either alone or in combination with chemical compounds, has been used for its therapeutic and antimicrobial effects. Photodynamic therapy encompasses the simultaneous action of a light source and photosensitizing agent in the presence of oxygen in tissues. Individually, each of these substances is innocuous, but their interaction is capable of giving rise to cytotoxic species that lead to cell death.The advantage of this approach is the avoidance of the development of resistance on the part of the target bacteria and damage to the adjacent tissues, since the antimicrobial effect is confined to the area covered by the dye and irradiated by the light, acting quickly on the target organisms. The efficacy of photodynamic therapy depends on the energy dose and output power employed.

Evaluation of degree of halitosis:

The portable Oral ChromaTM device (Abilit, Japan) will be employed. This device uses a highly sensitive gas semiconductor sensor.It will be connected to the computer with a specific software program that allows the creation of a graph corresponding to the peaks and concentrations of gases, measuring the VSC thresholds (0 to 1000 ppb), with considerable precision after eight minutes.

Analysis of volatile sulfur compounds:

* Hydrogen sulfide: values greater than 112 ppb indicate halitosis (SH2 ≥ 112 ppb);
* Methyl mercaptan: values greater than 26 ppb indicate halitosis (CH3SH ≥ 26 ppb);

A quantitative, controlled, cross-sectional, clinical trial will be carried out involving 130 teenagers. All individuals will be submitted to evaluations with Oral ChromaTM for the diagnosis of halitosis (scores SH2 ≥ 112 ppb and CH3SH ≥ 26 ppb) at the beginning of the study. Three post-treatment evaluations will be carried out: one hour, 24 hours and one week after treatment. The subjects selected will be randomly allocated to five groups:

1. Group 1 will receive treatment with a tongue scraper;
2. Group 2 and 3will receive photodynamic therapy applied to the posterior two thirds of the dorsum of the tongue;
3. Groups 4 and 5 will receive combined treatment (tongue scraper and photodynamic therapy).

The statistical analysis will include the chi-square test and Fisher's Exact Test. The Student's t-test and analysis of variance (ANOVA) will be used for the comparison of means. Pearson's correlation coefficients will be calculated to determine the strength of correlations between continuous variables. A 95% significance level will be considered on all statistical tests (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Signed statement of informed consent;
* Authorization by legal guardian for the diagnosis and treatment of halitosis (Appendix 2);
* Halitosis score using cysteine: S2H ≥ 112 ppb and/or CH3SH ≥ 26 ppb (Oral ChromaTM).

Exclusion Criteria:

* Dental-facial anomalies;
* Currently undergoing orthodontic and/or orthopedic treatment;
* Use of removable appliance, implant or denture;
* Periodontal disease;
* Teeth with carious lesions;
* Currently undergoing cancer treatment;
* History of antibiotic treatment in previous month;
* Pregnancy;
* Hypersensitivity to the photosensitizing agent employed.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 130 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Halitosis Scores | Prior to the initial photodynamic therapy on day 1 and 1, 24 and 168 hours post-photodynamic therapy
  It will be compare de score of voalitile sulfur compounds in parts per billion (ppb) of hydrogen sulfide (H2S) and methyl mercaptan (CH3SH3).

SECONDARY OUTCOMES:
Microbiological Analysis | Prior to the initial photodynamic therapy on day 1 and 1 and 24 hours post-photodynamic therapy
  Microbiological analyses of coated tongue will be performed before and after treatment using a 1-μl inoculation loop for the collection of biofilm samples from the dorsum of the tongue. The samples will be transferred to 1.5-ml vials with reduced transport fluid and placed in a vortex mixer for approximately 30 seconds for homogenization. Ten-fold serial dilution will be prepared in 180 μl of sterile phosphate buffered saline and aliquots of 10-2, 10-3, 10-4 and 10-5 will be transferred to plates with brain heart infusion agar. As the main bacteria responsible for the production of VSCs are Gram-negative, the plates will be incubated in anaerobic jar for 72 h at 37 °C, following by the quantification of colony-forming units (CFUs)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra K Bussadori, phd, Study Director — University of Nove de Julho; Rubia G Lopes, master, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, SP, São Paulo, Brazil

REFERENCES:
- [Derived] Costa da Mota AC, Franca CM, Prates R, Deana AM, Costa Santos L, Lopes Garcia R, Leal Goncalves ML, Mesquita Ferrari RA, Porta Santos Fernandes K, Kalil Bussadori S. Effect of photodynamic therapy for the treatment of halitosis in adolescents - a controlled, microbiological, clinical trial. J Biophotonics. 2016 Dec;9(11-12):1337-1343. doi: 10.1002/jbio.201600067. Epub 2016 Jun 1. PMID 27248838
- [Derived] Lopes RG, da Mota AC, Soares C, Tarzia O, Deana AM, Prates RA, Franca CM, Fernandes KP, Ferrari RA, Bussadori SK. Immediate results of photodynamic therapy for the treatment of halitosis in adolescents: a randomized, controlled, clinical trial. Lasers Med Sci. 2016 Jan;31(1):41-7. doi: 10.1007/s10103-015-1822-6. Epub 2015 Oct 28. PMID 26510574
- [Derived] Lopes RG, de Godoy CH, Deana AM, de Santi ME, Prates RA, Franca CM, Fernandes KP, Mesquita-Ferrari RA, Bussadori SK. Photodynamic therapy as a novel treatment for halitosis in adolescents: study protocol for a randomized controlled trial. Trials. 2014 Nov 14;15:443. doi: 10.1186/1745-6215-15-443. PMID 25394474